CLINICAL TRIAL: NCT02023541
Title: A Phase I Study of Proton Beam Therapy in the Treatment of Esophageal Cancer
Brief Title: Proton Beam Therapy to Treat Esophageal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of insurance coverage for proton beam treatment
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201310084
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resectable disease (Other): Patients with resectable disease will undergo treatment with proton beam therapy.
  Interventions: Radiation: Proton beam therapy
- Unresectable disease (Other): Patients with unresectable disease will undergo treatment with proton beam therapy.
  Interventions: Radiation: Proton beam therapy

INTERVENTIONS:
Radiation: Proton beam therapy

SUMMARY:
Assess progression-free survival and overall survival of proton beam therapy (PBT) for patients with resectable vs. unresectable esophageal cancer, and to assess patient-reported outcomes of PBT for esophageal cancer at 6 months following chemoradiation and physician-reported toxicity of PBT for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma or squamous cell carcinoma of the cervical or thoracic esophagus or gastroesophageal junction or cardia of stomach.
* Staged by PET/CT and esophagogastroduodenoscopy (EGD) OR CT w/contrast and EGD to have stage II or III disease. Endoscopic ultrasound (EUS) is encouraged but not required.
* Prior endoscopic mucosal resection (EMR) with a diagnosis of stage II or III esophageal cancer is eligible, irrespective of margin status.
* Induction chemotherapy prior to concurrent chemoradiation is allowed.
* Prior thoracic radiation is allowable if degree of overlap with the esophageal radiotherapy treatment is deemed to be safe by the treating radiation oncologist.
* At least 18 years of age.
* ECOG performance status ≤ 2 (Karnofsky > 60%)
* Normal bone marrow and organ function as defined below:

  * WBC > 2,500/mcL
  * Platelets ≥ 75,000/mcl
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤1.5 x IULN OR creatinine clearance ≥ 50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.
* English speaker.
* Financial coverage for proton therapy.

Exclusion Criteria:

* Planned treatment with radiation therapy alone without concurrent chemotherapy or chemotherapy alone.
* Previous or concomitant cancers within the past 3 years other than curatively treated carcinoma in situ of the cervix, basal cell carcinoma of the skin, curative treatment for transitional cell carcinoma of the bladder, and low risk prostate cancer. Except for prostate cancer (which can be observed if low risk), other cancers listed must have been treated in the past 3 years without evidence of recurrence at the time of registration.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia not controlled by pacer device, myocardial infarction within 3 months of registration, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 7 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 5 years
  Assess progression-free survival (PFS) of PBT for patients with resectable vs. unresectable esophageal cancer.
  PFS will be assessed using the Kaplan-Meier estimate.
Overall survival | 5 years
  Assess overall survival (OS) of PBT for patients with resectable vs. unresectable esophageal cancer.
  OS will be assessed using the Kaplan-Meier estimate.
Progression-free survival | 2 years
  Assess progression-free survival (PFS) of PBT for patients with resectable vs. unresectable esophageal cancer.
  PFS will be assessed using the Kaplan-Meier estimate.
Overall survival | 2 years
  Assess overall survival (OS) of PBT for patients with resectable vs. unresectable esophageal cancer.
  OS will be assessed using the Kaplan-Meier estimate.

SECONDARY OUTCOMES:
Patient-reported outcomes of PBT for esophageal cancer at 12 months following chemoradiation. | 1 year
  We will calculate descriptive statistics (mean, standard deviation, etc.) for all QOL data (EQ-5D, SF-12) in addition to other PROs (depressive symptoms, social support) at each evaluation period. Univariate tests will explore the associations among QOL and PROs using analysis of variance (ANOVA) and Fisher's exact test for correlation. Changes over time in QOL and PROs will be analyzed utilizing repeated-measures modeling techniques (repeated measures analysis of covariance).
Quality of life | 6 months
  Patient-reported outcomes of proton beam therapy (PBT) for esophageal cancer at 6 months following chemoradiation
  We will calculate descriptive statistics (mean, standard deviation, etc.) for all QOL data (EQ-5D, SF-12) in addition to other PROs (depressive symptoms, social support) at each evaluation period. Univariate tests will explore the associations among QOL and PROs using analysis of variance (ANOVA) and Fisher's exact test for correlation. Changes over time in QOL and PROs will be analyzed utilizing repeated-measures modeling techniques (repeated measures analysis of covariance).
Toxicity | 1 year
  We will compare the proportion of ≥Grade 3 gastrointestinal or pulmonary toxicity events against historical controls utilizing Binomial tests for proportion.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bradley, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu